CLINICAL TRIAL: NCT00715130
Title: Move and Moderate in Balance (MOVE'M): A TREC Worksite Health Study
Brief Title: Move and Moderate in Balance
Acronym: MOVE'M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Shirley A.A. Beresford, PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHCRC-6334; U54CA116847 (NIH)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Overweight; Obesity; Sedentary
Keywords: Energy; Obesity; Energy Balance; Physical Activity; Dietary Intake; Overweight; Sedentary; Worksite; Body Mass Index; Weight Maintenance
MeSH Terms: conditions — Overweight; Obesity; Sedentary Behavior; Motor Activity | interventions — Eating; Energy Metabolism; Energy Intake; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Energy Balance — We propose to develop and test a comprehensive intervention that will provide simple strategies related to dietary intake and energy expenditure that individuals can follow to achieve a balance in their energy intake and expenditure, while simultaneously changing structural and environmental cues to focus on promoting information, social support and opportunities for managing energy intake and increasing physical activity.
  Other Names: dietary intake; energy expenditure; energy intake; physical activity

SUMMARY:
H1: The increase in body mass index between baseline and two year follow-up among intervention worksites will be lower than that among control worksites, such that the differential change will be negative on average.

DETAILED DESCRIPTION:
Our overall objective is to develop and evaluate an intervention that will maintain or decrease body mass index; specifically, we will recruit and randomize 30 worksites to a two year intervention in which we will:

* Influence the worksite environment, including policies and procedures, by increasing worksite access to healthy foods and physical activity opportunities
* Promote individual behavior change, through increasing awareness of energy balance; building a physical activity intervention that will promote increased levels of energy expenditure through the combination of increased daily physical activity and regular, structured exercise; and building a dietary intervention that will promote decreased calorie intake.

Our primary aim is to:

1) Evaluate the effectiveness of the intervention in reducing or maintaining body mass index in a randomized controlled trial of worksites.

Our secondary aims are to:

1. Assess changes in worksite environment in access to healthy foods and physical activity opportunities attributable to the intervention
2. Assess changes in individual level physical activity and energy intake attributable to the intervention
3. Assess the changes in sequalae of weight loss including biomarkers of metabolic effects, and weight loss quality of life and symptom measures; and
4. Estimate the cost-effectiveness of the intervention in controlling weight.

ELIGIBILITY:
Inclusion Criteria:

* Employees of the enrolled worksite who are 18 years or older and work at the company at least 50% FTE (20 hrs per week)

Exclusion Criteria:

* Any employees of the enrolled worksite who are interns or seasonal workers or employees who work less than 50% FTE (20 hrs per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Our main outcome measure is change in body mass index, as an aggregated value at the worksite level. | At study conclusion

SECONDARY OUTCOMES:
Secondary, process measures will be of physical activity, physical fitness and calorie intake, at the individual level, within worksites. | At study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Shirley AA Beresford, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Anne McTiernan, MD, PhD, Study Director — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States